CLINICAL TRIAL: NCT01845350
Title: Safety and Feasibility of Autologous M2 Macrophage Transplantation in Treatment of Non-Acute Stroke Patients
Brief Title: Safety of Autologous M2 Macrophage in Treatment of Non-Acute Stroke Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Siberian Branch of the Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ekaterina Y. Shevela, Senior Researcher, Laboratory of Cellular Therapy, Research Institute of Clinical Immunology, Siberian Branch of the Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STR-M2-2013
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- M2 macrophages (Other): M2 macrophage introduction
  Interventions: Other: M2 macrophage introduction

INTERVENTIONS:
Other: M2 macrophage introduction — * Generation of autologous M2 macrophages from peripheral blood of non-acute stroke patients
  * Intrathecal introduction of autologous M2 macrophages

SUMMARY:
The purpose of this study is to determine whether M2 macrophages are safe and feasible in the treatment of non-acute stroke patients

DETAILED DESCRIPTION:
Our primary hypothesis is that autologous M2 macrophage transplantation via intrathecal introduction is feasible and safe after non-acute stroke. Our secondary hypothesis is that autologous M2 macrophage transplantation is associated with improved neurological outcome after non-acute stroke

ELIGIBILITY:
Inclusion Criteria:

* Computed tomography confirmed ischemic or hemorrhagic stroke
* Duration since stroke onset more than 3 and less than 12 months
* Age between 18 and 75 years old
* Persistent neurological deficits more than 4 points in NIHSS stroke scale
* Signed informed consent

Exclusion Criteria:

* The history of previous stroke
* Seizures
* Thrombophilias or primary hematological diseases
* Malignancy
* Hepatic or renal dysfunctions
* Hemodynamic or respiratory instability
* Autoimmune disease
* HIV or uncontrolled bacterial, fungal, or viral infections
* Pregnancy
* Participation in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The number of patients with severe adverse events | 1-3 days, 6 months
  Occurence of severe adverse events including mortality, neurological worsening and seizures

SECONDARY OUTCOMES:
Improvement of functional outcome in National Institutes of Health Stroke Scale (NIHSS) | 1-3 days, 6 months
Improvement in Barthel Index | 1-3 days, 6 months
Improvement in modified Rankin scale | 1-3 days, 6 months

OTHER OUTCOMES:
Number of patients with recurrent vascular episodes | 1-3 days, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena R. Chernykh, MD, PhD, Study Chair — Research Institute of Clinical Immunology, Russian Academy of Medical Sciences (Siberian Branch)
Locations (1):
- Research Institute of Clinical Immunology, Russian Academy of Medical Sciences (Siberian Branch), Novosibirsk, Russia

REFERENCES:
- [Result] Chernykh ER, Shevela EY, Starostina NM, Morozov SA, Davydova MN, Menyaeva EV, Ostanin AA. Safety and Therapeutic Potential of M2 Macrophages in Stroke Treatment. Cell Transplant. 2016;25(8):1461-71. doi: 10.3727/096368915X690279. Epub 2015 Dec 14. PMID 26671426